CLINICAL TRIAL: NCT04577469
Title: Randomized,One-period,Single Oral Dose,Open-label,Parallel,Bioequivalence Study to Compare 500mg Sulfadoxine/25mg Pyrimethamine Tablet Versus G-COSPE® Tablet (500mg Sulfadoxine/25mg Pyrimethamine) in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Sulfadoxine/ Pyrimethamine Tablets in Healthy Subjects Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Emzor Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 827-2018
Record Dates: First submitted 2020-02-26; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500 mg sulfadoxine / 25 mg pyrimethamine tablet (Experimental): 500 mg sulfadoxine / 25 mg pyrimethamine tablet will be administered once.
  Interventions: Drug: Maldox tablets; Drug: G-COSPE® tablets
- G-COSPE® tablets (Active Comparator): G-COSPE® tablets (500 mg sulfadoxine / 25 mg pyrimethamine) will be administered once.
  Interventions: Drug: Maldox tablets; Drug: G-COSPE® tablets

INTERVENTIONS:
Drug: Maldox tablets — 500 mg sulfadoxine / 25 mg pyrimethamine to be given as single dose once under fasting condition
Drug: G-COSPE® tablets — 500 mg sulfadoxine / 25 mg pyrimethamine to be given as single dose once under fasting condition

SUMMARY:
To asses bio equivalence between two (500 mg sulfadoxine / 25 mg pyrimethamine) formulation.

DETAILED DESCRIPTION:
The aim of this study is to assess bioequivalence between a single dose from the test product, Sulfadoxine/ Pyrimethamine tablets (500 mg sulfadoxine / 25 mg pyrimethamine), manufactured by Ms. Emzor Pharmaceuticals Industries Ltd, Nigeria versus the reference product G-COSPE® tablets (500 mg sulfadoxine / 25 mg pyrimethamine) manufactured by Guilin Pharmaceutical Co. Ltd, China under fasting conditions and to monitor the safety of the subjects.

ELIGIBILITY:
Inclusion criteria:

1. The subject is aged between eighteen & fifty years (18 - 50).
2. The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
3. The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
4. Results of medical history, vital signs, physical examination & conducted medical laboratory tests are normal as determined by the clinical investigator.
5. The subject tested negative for hepatitis (B & C) viruses and human immunodeficiency virus (HIV).
6. There is no history or evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
7. The subject is able to understand and willing to sign the informed consent form.
8. The subject has normal liver (AST & ALT enzymes) function.
9. The subject's kidney function tests are within normal ranges.
10. The subject has normal respiratory system.
11. The subject has normal platelet levels.
12. For female subjects: negative pregnancy test and the woman is using two reliable contraception methods.
13. The subject has normal cardiovascular system, ECG recording & QTc interval less than 450 ms.

Exclusion criteria:

1. The subject is a heavy smoker (more than 10 cigarettes per day).
2. The subject has suffered an acute illness one week before dosing.
3. The subject has a history of or concurrent consumption of alcohol.
4. The subject has a history of or concurrent consumption of illicit drugs.
5. The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
6. Subject who has been hospitalized within three months before the study or during the study.
7. Subject who is vegetarian.
8. The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 23 hours after dosing.
9. The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing and any time during the study, unless otherwise judged acceptable by the clinical investigator.
10. The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
11. The subjects who have been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study
12. The subjects who have donated blood within 80 days before first dosing.
13. The subject has a history presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Peak Plasma Concentration (Cmax) for Sulfadoxine and Pyrimethamine. | 12 weeks
  The average bioequivalence of the products will be concluded if the two-sided 90 % confidence interval for the test to reference ratio of the population means is within 80.00 - 125.00 % for the ln transformed data Cmax of sulfadoxine & pyrimethamine
Area under the plasma concentration versus time curves (AUC0 - 72) for Sulfadoxine and Pyrimethamine. | 12 weeks
  The average bioequivalence of the products will be concluded if the two-sided 90 % confidence interval for the test to reference ratio of the population means is within 80.00 - 125.00 % for the ln transformed data AUC0 -72 of sulfadoxine & pyrimethamine

SECONDARY OUTCOMES:
Obtaining the Tmax (Time to reach maximum concentration) for Sulfadoxine and Pyrimethamine | 12 weeks
  The descriptive statistics including Maximum, Minimum and Median values will be measured for Tmax.
ECG QTc Interval (safety and tolerability) | ECG recording will be performed 4 hours post- dosing and at the end of the study (at 72.00 hours post dosing) as follow-up tests
  Clinically significant abnormal deviations in ECG QTc interval
Blood pressure (safety and tolerability) | At 1-hour pre-dosing; 2, 4, 6, 8, 12 and 23 hours post-dosing (±45 minutes of scheduled time). Blood pressure will also be measured at 48 and 72 hours post-dosing upon ambulatory sample collection.
  Clinically significant abnormal deviations. Normal range of blood pressure > 90/60 and <140/90 mmHg. Treatment will be offered to those subjects whom blood pressure drops to 90/60 mm Hg or less and the subject will be excluded in case of not responding to treatment.
Pulse (safety and tolerability) | At 1-hour pre-dosing; 2, 4, 6, 8, 12 and 23 hours post-dosing (±45 minutes of scheduled time). Pulse will also be measured at 48 and 72 hours post-dosing upon ambulatory sample collection.
  Clinically significant abnormal deviations. Normal range of Pulse 60-100 Bpm.
Temperature (safety and tolerability) | At 1-hour pre-dosing; 2, 6, 10, 14, 18, 22 & 23 hours post-dosing (±45 minutes of scheduled time). Temperature will also be measured at 48 and 72 hours post-dosing upon ambulatory sample.
  Clinically significant abnormal deviations. The temperature will be measured axillary, orally or using infrared thermometer, standardized across all subjects. Normal range of temperature 36.5-37.5 ºC.
Respiratory rate (safety and tolerability) | At 1-hour pre-dosing; 2, 6, 10, 14, 18, 22 & 23 hours post-dosing (±45 minutes of scheduled time). Respiratory rate will also be measured at 48 and 72 hours post-dosing upon ambulatory sample.
  Clinically significant abnormal deviations. Normal range of respiratory rate 12-18 B/M
Hematology (Safety and Tolerability) | At the end of the study (at 72.00 hours post dosing)
  Hematology test will include Complete blood count
Number of Subjects With AEs | At 12 and 1-hour pre-dosing; 2, 4, 6, 8, 10, 12, 23, 48 and 72 hours post-dosing
  Safety and tolerability: number of subjects with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Abu Fara, MD,Internist, Principal Investigator — ACDIMA Biocenter

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ICH E6(R2) guideline — https://www.ema.europa.eu/en/documents/scientific-guideline/ich-e-6-r2-guideline-good-clinical-practice-step-5_en.pdf